CLINICAL TRIAL: NCT04520243
Title: Evaluation of Letters Versus Numbers (ELEVEN) Study: ETDRS Visual Acuity Chart Performance in an English Alphabet Illiterate Population
Brief Title: Evaluation of Letters Versus Numbers (ELEVEN) Study
Acronym: ELEVEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Nicholas Fung, Clinical Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ELEVEN
Record Dates: First submitted 2020-08-17; First posted 2020-08-20 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Visual Acuity
Keywords: ETDRS visual acuity; English alphabet illiterate; ETDRS number chart

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- English alphabet illiterate group (Experimental): Individuals with no self-reported understanding of English alphabet and recognition of <6/10 Sloan Letters
  Interventions: Diagnostic Test: Visual acuity assessment by ETDRS charts
- English alphabet literate group (Active Comparator): Individuals with self-reported understanding of English alphabet and recognition of ≥6/10 Sloan Letters
  Interventions: Diagnostic Test: Visual acuity assessment by ETDRS charts

INTERVENTIONS:
Diagnostic Test: Visual acuity assessment by ETDRS charts — All participants must complete VA measurement of both eyes using 2 charts including the ETDRS letters chart and ETDRS numbers chart.

SUMMARY:
This is a prospective randomised controlled trial to determine the performance of Best Corrected Visual Acuity (BCVA) scores using the ETDRS number chart were compared with ETDRS alphabet chart in healthy eyes of patients who do not recognise the English alphabet.

DETAILED DESCRIPTION:
BACKGROUND: The measurement of visual acuity is important in the clinical setting to assess visual function and treatment response, while in research to provide objective clinical outcomes. The current gold standard for visual acuity measurement in most research studies, including major clinical trials, is the Early Treatment Diabetic Retinopathy Study (ETDRS) chart designed by Bailey and Lovie. However, this may not be suitable for participants who are illiterate. Alternatives exist, including the ETDRS numbers chart, Landolt C chart and Tumbling E chart. Existing studies show that the Landolt C and Tumbling E charts are alternatives with agreement with ETDRS letters chart in healthy and diseased eyes. However, the charts are limited by their 25% (if four orientations) or 12.5% (if eight orientations) chance of guessing the orientation of the letter.

The ETDRS numbers chart may overcome this limitation, as it uses five unique numbers instead of a single rotating letter. There are few studies evaluating the different types of visual acuity measurement among those unfamiliar with the English alphabet. Though one study shows high repeatability and agreement between the ETDRS letters and numbers charts in healthy and diseased eyes of English literate individuals and shorter testing duration when using the numbers chart, this finding has not been validated in individuals unfamiliar with the English alphabet. This study aims to evaluate how the ETDRS letters and numbers charts compare in individuals unfamiliar with the English alphabet.

METHODS: Eligible subjects were divided into 2 groups according to level of literacy. Literacy was determined by self-reported exposure to the English alphabet and recognition of the 10 Sloan letters (C, D, H, K, N, O, R, S, V, and Z). Subjects included were classified into the 2 groups: group A, with no exposure to the English alphabet and recognition of <6/10 letters, and group B, with exposure to the English alphabet and recognition of ≥6/10 letters.

Testing: Each subject underwent 2 rounds of BCVA measurements using 2 types of ETDRS charts in randomized sequence as follows: LN or NL (L = ETDRS letters chart, N = ETDRS numbers chart) from Precision Vision® (PV). The randomization of the testing sequence was performed by a study coordinator independent of study recruiter, optometrist or investigator. Sequentially numbered, opaque and sealed envelopes were used for allocation concealment and opened by the optometrist prior to testing.

The tests were performed and recorded by a single optometrist in the same testing room with similar lighting conditions. For every round of testing, the right eye was examined first, followed by the left eye. For the right eye, numbers chart (PV No. 2702A) and letters chart (PV No. 2173) were used. For the left eye, the numbers chart (PV No. 2714A) and letters chart (PV No. 2174) were used. Different charts (with the same optotypes but in different order) were used for right and left eyes to minimize the effect of learning between consecutive tests.

ELIGIBILITY:
Inclusion Criteria:

1. Hong Kong residents
2. Age 50 years or above
3. Attending Southern District Screening program

Exclusion Criteria:

1. BCVA 20/200 or below
2. Any clinically relevant ocular disease that might affect visual acuity

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
BCVA Measurements | 1 day
  Assessment of BCVA using ETDRS numbers and letters chart and its comparison between the testing groups and intervention methods. All visual acuity tests were performed at 3 metres with at least 15 seconds between each chart. Subjects were asked to read as many optotypes as possible according to the ICO Visual Acuity Measurement Standard.
Testing Duration | 1 day
  Assessment of testing duration using ETDRS numbers and letters and its comparison between the testing groups and intervention methods. The testing durations of each visual acuity test were measured and recorded by a single timekeeper with a standard digital chronometer.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Fung, Principal Investigator — Department of Ophthalmology, HKU
Locations (1):
- HKSDS Program, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
By request to corresponding users
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Within 1 year of publication
Access Criteria: For research publisher

REFERENCES:
- [Background] Bailey IL, Lovie JE. New design principles for visual acuity letter charts. Am J Optom Physiol Opt. 1976 Nov;53(11):740-5. doi: 10.1097/00006324-197611000-00006. PMID 998716
- [Background] Ferris FL 3rd, Bailey I. Standardizing the measurement of visual acuity for clinical research studies: Guidelines from the Eye Care Technology Forum. Ophthalmology. 1996 Jan;103(1):181-2. doi: 10.1016/s0161-6420(96)30742-2. No abstract available. PMID 8628551
- [Background] Kniestedt C, Stamper RL. Visual acuity and its measurement. Ophthalmol Clin North Am. 2003 Jun;16(2):155-70, v. doi: 10.1016/s0896-1549(03)00013-0. PMID 12809155
- [Background] Chaikitmongkol V, Nanegrungsunk O, Patikulsila D, Ruamviboonsuk P, Bressler NM. Repeatability and Agreement of Visual Acuity Using the ETDRS Number Chart, Landolt C Chart, or ETDRS Alphabet Chart in Eyes With or Without Sight-Threatening Diseases. JAMA Ophthalmol. 2018 Mar 1;136(3):286-290. doi: 10.1001/jamaophthalmol.2017.6290. PMID 29346499
- [Background] Koenig S, Tonagel F, Schiefer U, Bach M, Heinrich SP. Assessing visual acuity across five disease types: ETDRS charts are faster with clinical outcome comparable to Landolt Cs. Graefes Arch Clin Exp Ophthalmol. 2014 Jul;252(7):1093-9. doi: 10.1007/s00417-014-2670-y. Epub 2014 May 28. PMID 24867313
- [Background] Treacy MP, Hurst TP, Conway M, Duignan ES, Dimitrov BD, Brennan N, Cassidy L. The early treatment in diabetic retinopathy study chart compared with the tumbling-E and Landolt-C. Ophthalmology. 2015 May;122(5):1062-3.e1. doi: 10.1016/j.ophtha.2014.11.024. Epub 2015 Jan 10. No abstract available. PMID 25582784
- [Background] Kuo HK, Kuo MT, Tiong IS, Wu PC, Chen YJ, Chen CH. Visual acuity as measured with Landolt C chart and Early Treatment of Diabetic Retinopathy Study (ETDRS) chart. Graefes Arch Clin Exp Ophthalmol. 2011 Apr;249(4):601-5. doi: 10.1007/s00417-010-1461-3. Epub 2010 Jul 24. PMID 20658145
- [Background] Ruamviboonsuk P, Tiensuwan M, Kunawut C, Masayaanon P. Repeatability of an automated Landolt C test, compared with the early treatment of diabetic retinopathy study (ETDRS) chart testing. Am J Ophthalmol. 2003 Oct;136(4):662-9. doi: 10.1016/s0002-9394(03)00394-5. PMID 14516806
- [Background] Doig GS, Simpson F. Randomization and allocation concealment: a practical guide for researchers. J Crit Care. 2005 Jun;20(2):187-91; discussion 191-3. doi: 10.1016/j.jcrc.2005.04.005. PMID 16139163
- [Background] Universal C: Visual Acuity Measurement Standard. Visual Functions Committee 1984.